# Proefpersoneninformatie voor deelname aan medisch-wetenschappelijk onderzoek

Tijd in de acute zorgketen (Time within the Acute Care Chain 2 – TACC 2 trial)

# **Inleiding**

Geachte heer/mevrouw,

Wij vragen u om mee te doen aan een medisch-wetenschappelijk onderzoek. Meedoen is vrijwillig. Om mee te doen is wel uw schriftelijke toestemming nodig. U ontvangt deze brief omdat u op de spoedeisende hulp (SEH) behandeld wordt en daarmee in aanmerking komt voor het onderzoek. Dit onderzoek zal plaatsvinden op de SEH in Heerlen. Aan dit onderzoek zullen naar verwachting 750 proefpersonen meedoen.

Dit onderzoek is beoordeeld door de Medisch Ethische Toets Commissie Zuyd (METC-Z).

Voordat u beslist of u wilt meedoen aan dit onderzoek, krijgt u uitleg over wat het onderzoek inhoudt. Lees deze informatie rustig door en vraag de onderzoeker uitleg als u vragen heeft. U kunt er ook over praten met uw partner, vrienden of familie.

## 1. Doel van het onderzoek

Op de SEH komen mensen met veel verschillende aandoeningen, meestal na een verwijzing van de huisarts, of nadat de ambulance medewerker de patiënt thuis onderzocht heeft. Het is niet bekend hoe lang het traject is dat patiënten ondergaan voordat ze op de SEH terecht komen (dus vanaf het moment dat u vandaag contact zocht met een hulpverlener tot en met behandeling op de SEH). Met dit onderzoek willen we dat onderzoeken.

#### 2. Wat meedoen inhoudt

Meedoen aan dit onderzoek houdt in dat u samen met uw naasten en de onderzoeker een korte vragenlijst (enkele minuten) invult over de duur van het traject voorafgaand aan uw SEH-bezoek vandaag. Deze vragenlijst wordt op papier ingevuld tijdens het SEH bezoek. Zo nodig raadpleegt de onderzoeker uw dossier om vragen die u niet direct kunt beantwoorden toch in te kunnen vullen. Denk hierbij bijvoorbeeld aan de (voorlopige) diagnose die de arts vandaag stelt / gesteld heeft, of het exacte tijdstip dat u op de SEH aankwam.

Uw behandeling vandaag wordt niet beïnvloed door uw beslissing of u wel of niet deelneemt aan het onderzoek.

Het onderzoek is ten einde op het moment dat u de SEH verlaat.

## 3. Wat wordt er van u verwacht

Om het onderzoek goed te laten verlopen is het belangrijk dat u zich aan de volgende afspraken houdt. De afspraken zijn dat u:

- de instructies van de onderzoeker volgt
- het aan de onderzoeker meldt als u ook nog aan een ander medisch-wetenschappelijk onderzoek meedoet/wil meedoen

Het is belangrijk dat u contact opneemt met de onderzoeker als:

- u niet meer wilt meedoen aan het onderzoek
- uw contactgegevens wijzigen

# 4. Mogelijke voor- en nadelen

Bij dit onderzoek zijn de risico's die u loopt bij deelname nagenoeg nihil. Het is wel belangrijk dat u de mogelijke voor- en nadelen goed afweegt voordat u besluit mee te doen. De voordelen van meedoen aan het onderzoek zijn voornamelijk de verbetering van zorg voor patiënten zoals u op de langere termijn. Eventuele nadelen zijn nihil. Wij zijn u dankbaar voor uw tijdsinvestering in het onderzoek mocht u besluiten mee te willen doen.

# 5. Als u niet wilt meedoen of wilt stoppen met het onderzoek

U beslist zelf of u meedoet aan het onderzoek. Deelname is vrijwillig. Als u besluit niet mee te doen, hoeft u verder niets te doen. U hoeft niets te tekenen. U hoeft ook niet te zeggen waarom u niet wilt meedoen. Als u patiënt bent wordt u op de gebruikelijke manier behandeld.

Als u wel meedoet, kunt u zich altijd bedenken en toch stoppen, ook tijdens het onderzoek. Als u patiënt bent dan wordt u weer op de gebruikelijke manier behandeld. U hoeft niet te zeggen waarom u stopt. Wel moet u dit direct melden aan de onderzoeker. De gegevens die tot dat moment zijn verzameld, worden gebruikt voor het onderzoek.

Als er nieuwe informatie over het onderzoek is die belangrijk voor u is, laat de onderzoeker dit aan u weten. U wordt dan gevraagd of u blijft meedoen.

#### 6. Einde van het onderzoek

Uw deelname aan het onderzoek stopt als:

- u uw bijdrage aan het onderzoek zoals hiervoor beschreven geleverd heeft
- u zelf kiest om te stoppen
- het einde van het hele onderzoek zoals hiervoor beschreven is bereikt
- de onderzoeker het beter voor u vindt om te stoppen
- de Raad van Bestuur, de overheid of de beoordelende medisch-ethische toetsingscommissie besluit om het onderzoek te stoppen

## 7. Gebruik en bewaren van uw gegevens

Voor dit onderzoek worden uw persoonsgegevens verzameld, gebruikt en bewaard. Het gaat om gegevens zoals uw naam, adres, geboortedatum en om gegevens over uw gezondheid. Het verzamelen, gebruiken en bewaren van uw gegevens is nodig om de vragen die in dit onderzoek worden gesteld te kunnen beantwoorden en de resultaten te kunnen publiceren. Wij vragen voor het gebruik van uw gegevens uw toestemming.

# Vertrouwelijkheid van uw gegevens

Om uw privacy te beschermen krijgen uw gegevens een code. Uw naam en andere gegevens die u direct kunnen identificeren worden daarbij weggelaten. Alleen met de sleutel van de code zijn gegevens tot u te herleiden. De sleutel van de code blijft veilig opgeborgen in de lokale onderzoeksinstelling. Ook in rapporten en publicaties over het onderzoek zijn de gegevens niet tot u te herleiden.

## Toegang tot uw gegevens voor controle

Sommige personen kunnen op de onderzoekslocatie toegang krijgen tot al uw gegevens. Ook tot de gegevens zonder code. Dit is nodig om te kunnen controleren of het onderzoek goed en betrouwbaar is uitgevoerd. Personen die ter controle inzage krijgen in uw gegevens zijn nationale en internationale

toezichthoudende autoriteiten, bijvoorbeeld, de Inspectie Gezondheidszorg en Jeugd. Zij houden uw gegevens geheim. Wij vragen u voor deze inzage toestemming te geven.

## Bewaartermijn gegevens

Uw gegevens moeten 15 jaar worden bewaard op de onderzoekslocatie.

## Bewaren en gebruiken van gegevens

Uw gegevens kunnen na afloop van dit onderzoek ook nog van belang zijn voor ander wetenschappelijk onderzoek op het gebied van uw aandoening en/of van de verdere ontwikkeling van de acute zorg. Daarvoor zullen uw gegevens 15 jaar worden bewaard. U kunt op het toestemmingsformulier aangeven of u hier wel of niet mee instemt. Indien u hier niet mee instemt, kunt u gewoon deelnemen aan het huidige onderzoek.

#### Intrekken toestemming

U kunt uw toestemming voor gebruik van uw persoonsgegevens altijd weer intrekken. Dit geldt voor dit onderzoek en ook voor het bewaren en het gebruik voor het toekomstige onderzoek. De onderzoeksgegevens die zijn verzameld tot het moment dat u uw toestemming intrekt worden nog wel gebruikt in het onderzoek.

## Meer informatie over uw rechten bij verwerking van gegevens

Voor algemene informatie over uw rechten bij verwerking van uw persoonsgegevens kunt u de website van Zuyderland en de Autoriteit Persoonsgegevens raadplegen. Bij vragen over uw rechten kunt u contact opnemen met de verantwoordelijke voor de verwerking van de persoonsgegevens. Voor dit onderzoek is dat Drs. L. Claassen, SEH-arts KNMG. Zie bijlage A voor contactgegevens. Bij vragen of klachten over de verwerking van uw persoonsgegevens raden we u aan eerst contact op te nemen met de onderzoekslocatie. U kunt ook contact opnemen met de Functionaris voor de Gegevensbescherming van de instelling, zie bijlage A voor de contactgegevens, of de Autoriteit Persoonsgegevens.

# 8. Heeft u vragen of een klacht?

Bij vragen kunt u contact opnemen met het onderzoeksteam. Indien u klachten heeft over dit onderzoek, dan kunt u dit bespreken met de onderzoeker of uw behandelend arts. Wilt u dit liever niet, dan kunt u zich wenden tot de klachtenfunctionaris van Zuyderland. Alle gegevens vindt u in **bijlage A**: Contactgegevens.

## 9. Ondertekening toestemmingsformulier

Wanneer u voldoende bedenktijd heeft gehad, wordt u gevraagd te beslissen over deelname aan dit onderzoek. Indien u toestemming geeft, zullen wij u vragen deze op de bijbehorende toestemmingsverklaring schriftelijk te bevestigen. Door uw schriftelijke toestemming geeft u aan dat u de informatie heeft begrepen en instemt met deelname aan het onderzoek. Zowel uzelf als de onderzoeker ontvangen een getekende versie van deze toestemmingsverklaring.

Dank voor uw aandacht.

# Bijlagen bij deze informatie

- A. Contactgegevens
- B. Toestemmingsformulier

## Bijlage A: contactgegevens voor Zuyderland

## (Lokale) Hoofdonderzoeker

Naam: Drs. G. Latten Functie: SEH-arts KNMG

Contactgegevens: g.latten@zuyderland.nl

Bereikbaarheid: 088-4597777

## [Hoofdonderzoeke/coördinerende onderzoeker/uitvoerende onderzoeker]

Naam: Drs. L. Claassen Functie: SEH-arts KNMG

Contactgegevens: l.claassen@zuyderland.nl

Bereikbaarheid: 088-4597777

## Klachten

Indien u klachten heeft over het onderzoek, kunt u dit bespreken met de onderzoeker of uw behandelend arts. Wilt u dit liever niet, dan kunt u zich wenden tot een van de klachtenfunctionarissen van Zuyderland, e-mail: klachtenfunctionarisziekenhuis@zuyderland.nl, tel. 088-459 7603.

# Meer informatie over uw rechten bij verwerking van gegevens

Voor algemene informatie over uw rechten bij verwerking van uw persoonsgegevens kunt u de website van de Autoriteit Persoonsgegevens raadplegen. Bij vragen of klachten over het gebruik of de verwerking van uw gegevens, of over uw rechten, kunt u contact opnemen met:

# Functionaris Gegevensbescherming (FG) van Zuyderland Medisch Centrum ZIEKENHUIS/CURE

Naam: Marianne Korpershoek

Tel +31-88-4597777

E-mail: <a href="mailto:privacy@zuyderland.nl">privacy@zuyderland.nl</a>

Link naar website instelling met privacyverklaring/privacy reglement:

 $\underline{https://www.zuyderland.nl/wp-content/uploads/2016/06/Privacyreglement-t.b.v.-}$ 

patiëntgegevens.pdf

PIF - TACC trial

| Patientsticker + nummer |
|-------------------------|

# Bijlage B: toestemmingsformulier proefpersoon

# Tijd in de acute zorgketen (Time within the Acute Care Chain – TACC trial)

- Ik heb de informatiebrief gelezen. Ook kon ik vragen stellen. Mijn vragen zijn voldoende beantwoord. Ik had genoeg tijd om te beslissen of ik meedoe.
- Ik weet dat meedoen vrijwillig is. Ook weet ik dat ik op ieder moment kan beslissen om toch niet mee te doen of te stoppen met het onderzoek. Daarvoor hoef ik geen reden te geven.
- Ik geef toestemming voor het opvragen van informatie bij mijn huisarts.
- Ik geef toestemming voor het verzamelen en gebruiken van mijn gegevens voor de beantwoording van de onderzoeksvraag in dit onderzoek.
- Ik weet dat voor de controle van het onderzoek sommige mensen toegang tot al mijn gegevens kunnen krijgen. Die mensen staan vermeld in deze informatiebrief. Ik geef toestemming voor die inzage door deze personen.

| | Ik geef | □ wel |
|---|---|---|
| - | ik geei | □ geen toestemming om mijn persoonsgegevens langer te bewaren en te gebruiker voor toekomstig onderzoek op het gebied van mijn aandoening en/of van de verdere ontwikkeling van de acute zorg. |
| - | Ik geef | □ wel |
| | | □ <b>geen</b> toestemming om mij na dit onderzoek opnieuw te benaderen voor een vervolgonderzoek. |
| - | Ik wil mee | edoen aan dit onderzoek. |
| | am proefper<br>ndtekening: | rsoon: Datum :// |
| | | ik deze proefpersoon volledig heb geïnformeerd over het genoemde onderzoek. |
| | - | et onderzoek informatie bekend wordt die de toestemming van de proefpersoon zou<br>beden, dan breng ik hem/haar daarvan tijdig op de hoogte. |
| Naa | am onderzo | eker (of diens vertegenwoordiger): |
| Har | ndtekening: | Datum: / / |

\* Doorhalen wat niet van toepassing is.

De proefpersoon krijgt een volledige informatiebrief mee, samen met een kopie van het getekende toestemmingsformulier.